CLINICAL TRIAL: NCT05219383
Title: Clinical and Electrophysiological Patterns of Chronic Dysimmune Polyneuropathy Among Patients Attending Neuropsychiatry Department - Assiut University
Brief Title: Clinical and Electrophysiological Patterns of Chronic Dysimmune Polyneuropathy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yousef Josef Louis Megalla, principle investigator, Assiut University
Other Study IDs: Chronic dysimmune neuropathy
Record Dates: First submitted 2021-12-31; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic dysimmune neuropathies (CDN) are a heterogenous group of acquired inflammatory demyelinating neuropathies including chronic inflammatory demyelinating polyneuropathies (CIDP), Lewis-Sumner Syndrome (LSS), multifocal motor neuropathy (MMN) and other rare entities.

Despite their relatively low prevalence, CDN lead to substantial costs for patients and society. CDN are usually misdiagnosed due to progressive nature of the disease with little known data regarding disease activity and treatment response

DETAILED DESCRIPTION:
CIDP is the most common treatable CDN worldwide. Its prevalence is ranging between approximately 1 to 8.9 cases per 100.000 . In addition, there is often the tendency to diagnose CIDP in order to attempt a treatment option. This ultimately leads to overdiagnosis and overtreatment in some patients

Although the different CDN have varying underlying pathophysiology and clinical characteristics, they are all potentially treatable with immunomodulatory drugs.

To date, diagnostic criteria, measurement of disease activity and treatment response of CDN are mainly based on clinical, electrophysiological, and patient related outcome parameters. The commonly used EFNS/PNS diagnostic criteria for CIDP seems to have the best sensitivity among different sets of diagnostic criteria

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, both sexes, history of sensory and/or motor complaint with progressive course over more 2 months

Exclusion Criteria:

* *Patients with systemic diseases (DM, chronic kidney or liver disease, thyroid disease, vitamin B12 deficiency)

  * Family history of peripheral neuropathy or neurological symptoms suggestive for heredo-familial neurological disorders
  * Patients with infective cause as (HBV, HCV, HIV, leprosy)
  * Toxic and drug induced polyneuropathy (chemotherapeutics, antimicrobial ..

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age > 18 years, both sexes, history of sensory and/or motor complaint with progressive course over more 2 months
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients diagnosed with chronic inflammatory demyleinating polyneuropathy attending neuropsychiatry department Assiut university | From January 2023 to December 2026
  Number of patients diagnosed with chronic inflammatory demyleinating polyneuropathy attending neuropsychiatry department Assiut university

REFERENCES:
- [Background] Rajabally YA, Nicolas G, Pieret F, Bouche P, Van den Bergh PY. Validity of diagnostic criteria for chronic inflammatory demyelinating polyneuropathy: a multicentre European study. J Neurol Neurosurg Psychiatry. 2009 Dec;80(12):1364-8. doi: 10.1136/jnnp.2009.179358. Epub 2009 Jul 20. PMID 19622522
- [Background] Breiner A, Brannagan TH 3rd. Comparison of sensitivity and specificity among 15 criteria for chronic inflammatory demyelinating polyneuropathy. Muscle Nerve. 2014 Jul;50(1):40-6. doi: 10.1002/mus.24088. Epub 2013 Dec 11. PMID 24338746
- [Background] Hartung HP, Lehmann HC, Willison HJ. Peripheral neuropathies: Establishing common clinical research standards for CIDP. Nat Rev Neurol. 2011 May;7(5):250-1. doi: 10.1038/nrneurol.2011.46. Epub 2011 Apr 12. No abstract available. PMID 21537353